CLINICAL TRIAL: NCT05457595
Title: Phase II Clinical Study on the Re-irradiation of Lateral Pelvic Recurrences of Gynecological Malignancies
Brief Title: Clinical Study on the Re-irradiation of Lateral Pelvic Recurrences of Gynecological Malignancies
Acronym: CYCLOPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNAO 41 2020C
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Tumor Recurrence; Malignant Epithelial Neoplasm of Vulva; Malignant Epithelial Tumor of Ovary; Malignant Epithelial Neoplasm
Keywords: gynecological cancer; carbon ion radiation therapy; recurrencies; CIRT
MeSH Terms: conditions — Recurrence; Vulvar Neoplasms; Ovarian Neoplasms; Carcinoma | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will undergo to carbon ion radiation therapy. It is a monocentric, prospective II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- carbon ion radiotherapy (Experimental): All enrolled subjects will undergo carbon ion radiation therapy. Patients affected by pelvic recurrence of gynecological neoplasia, already undergone to radiotherapy on pelvis, will be enrolled in the study.
  Interventions: Radiation: carbon ion radiation therapy

INTERVENTIONS:
Radiation: carbon ion radiation therapy — CIRT: Planning Target Volume (PTV) will be delivered a total dose of 48-52.8 GyRBE in 12 fractions, 4 fractions per week. Treatment duration 3 weeks.
  Treatment lasting more than 5 weeks or cases of treatment with less than 6 fractions in 14 consecutive days will not be accepted.
  Other Names: CIRT

SUMMARY:
The study aims to obtain a local control rate in patients with lateral pelvic relapses of gynecologycal cancers previously irradiated. High LET (Linear Energy Transfer) particles as carbon ions can guarantee a biologic advantage compared to photons in radioresistant neoplasms, given to their higher biological efficacy (RBE).

DETAILED DESCRIPTION:
Primary aim: estimate the effect, in terms of clinical response, of carbon ion treatment (CIRT) in patients with lateral pelvic recurrences of gynecological malignancies.

Secondary aims:

1. To describe the safety profile of carbon ion therapy.
2. To estimate the effect, in terms of survival, of carbon ion treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Karnofsky Index ≥ 70
* Histological or radiological diagnosis of pelvic and groin recurrence
* Contraindications for radical surgery
* No other distant progression or stable disease (SD) of known secondarisms (≥6 months)
* Previous radiation therapy on pelvis
* Distance ≥ 10mm between tumour and close intestinal tract (small intestine), radiologically evaluated
* Possibility to perform a surgery to space the intestinal loops, in case of distance < 10mm
* If needed, spacer in biocompatible material (silicon, goretex) or anatomical material (omentum, muscle patch), non-absorbable.
* DICOM (Digital Imaging and COmmunications in Medicine) images of the previous treatment plan availability
* Written informed consent
* Patient's ability to understand the characteristics and consequences of the clinical trial

Exclusion Criteria:

* Hip prosthesis, metal prostheses or any other condition that prevents adequate imaging to identify the target volume and calculate the dose in the treatment plan

  * Intestinal infiltration
  * Bladder infiltration
  * Vessel infiltration
  * Previous therapy with anti-angiogenesis drugs
  * Psychic or other disorders that may prevent informed consent
  * Previous invasive tumor, with the exception of skin cancer (excluding melanoma) unless disease-free for at least 3 years
  * Spacer in absorbable material (i.e. vycril)
  * Distance < 10mm between tumour and close intestinal tract (small intestine), radiologically evaluated
  * Impossibility to assess MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The research applies to gynecological tumors.
Enrollment: 55 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2028-02-24 (Estimated); Study Completion 2028-02-25 (Estimated)

PRIMARY OUTCOMES:
local control | 1 year after treatment
  absence of progression disease, in patients with lateral pelvic recurrences of gynecological malignancies
complete response | 1 year after treatment
  complete regression of the tumor lesion
partial response | 1 year after treatment
  Reduction of the tumor volume > 65% of the initial volume
stable disease | 1 year after treatment
  Volume between PR and PD
progression disease | 1 year after treatment
  Volume increase > 73% of the initial volume.

SECONDARY OUTCOMES:
overall survival | 1 year after treatment
  overall survival
Toxicity assessment according to CTCAE v. 5 | 1 year after treatment
  Tto define acute, intermediate and late toxicities according to Common Terminology Criteria for Adverse Events (CTCAE version 5.0)
Progression free survival | 1 year after treatment
  Progression free survival (PFS) with qualitative evaluation as a narrative of progression

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Barcellini, MD, Principal Investigator — CNAO National Center of Oncological Hadrontherapy
Locations (1):
- CNAO, Pavia, Pv, Italy